CLINICAL TRIAL: NCT06905327
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered QCZ484 in Healthy Subjects and Subjects With Mild Hypertension
Brief Title: A Study to Evaluate the Safety of QCZ484 in Healthy and Mild Hypertensive Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CQCZ484A02101; BW-00163-1002 (Other: Argo Biopharma)
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Mild Hypertension
Keywords: Hypertension; QCZ484
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part A: QCZ484 50 mg (Experimental): Healthy Cohort: single dose
  Interventions: Drug: QCZ484
- Part A: QCZ484 150 mg (Experimental): Healthy Cohort: single dose
  Interventions: Drug: QCZ484
- Part A: QCZ484 300 mg (Experimental): Healthy Cohort: single dose
  Interventions: Drug: QCZ484
- Part A: QCZ484 600 mg (Experimental): Healthy Cohort: single dose
  Interventions: Drug: QCZ484
- Part A: QCZ484 Placebo (Placebo Comparator): Healthy Cohort: single dose
  Interventions: Drug: Placebo
- Part B: QCZ484 150 mg (Experimental): Hypertension Cohort: single dose
  Interventions: Drug: QCZ484
- Part B: QCZ484 300 mg (Experimental): Hypertension Cohort: single dose
  Interventions: Drug: QCZ484
- Part B: QCZ484 600 mg (Experimental): Hypertension Cohort: single dose
  Interventions: Drug: QCZ484
- Part B: QCZ484 Placebo (Placebo Comparator): Hypertension Cohort: single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QCZ484 — doses of 50, 150, 300 or 600 mg via subcutaneous injection
  Arms: Part A: QCZ484 150 mg; Part A: QCZ484 300 mg; Part A: QCZ484 50 mg; Part A: QCZ484 600 mg; Part B: QCZ484 150 mg; Part B: QCZ484 300 mg; Part B: QCZ484 600 mg
Drug: Placebo — via subcutaneous injection
  Arms: Part A: QCZ484 Placebo; Part B: QCZ484 Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study including Part A single ascending dose (SAD) in healthy subjects and Part B single dose in subjects with mild hypertension.

DETAILED DESCRIPTION:
Phase 1, multicenter, randomized, double-blind, placebo-controlled study to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of QCZ484. In Part A, single ascending doses of QCZ484 are tested in healthy subjects, while in Part B, single doses of QCZ484 are tested in subjects with mild hypertension. One dose of QCZ484 is administered subcutaneously.

This study was started by Argo Biopharma, and global sponsorship was transferred to Novartis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females aged 18 to 60 years, inclusive, at the time of informed consent. (Part A only).
* Males or females aged 18 to 72 years, inclusive, at the time of informed consent (Part B only).
* Body mass index (BMI) >= 18 and <= 32 kg/m2 and body weight >50 kg (Part A only).
* Body mass index (BMI) >=18 and <=35 kg/m2 and body weight >50 kg (Part B only).
* Triplicate 12-lead electrocardiogram (ECG) after >5 minutes resting without clinically significant findings at screening and Day -1.
* Mean sitting systolic blood pressure (SBP) of >=130 and <160 mm Hg (Part B only).

Exclusion Criteria:

* History of hypotension or orthostatic hypotension.
* History of syncope within 1 year.
* SBP <90 mmHg or DBP <60 mm Hg at screening (Part A only).
* Clinical laboratory findings outside of range are deemed clinically significant by the investigator at screening.
* Any liver function panel analyte value > 1.2 ×upper limits of normal (ULN) at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs) | Part A: up to 12 weeks post dose. Part B: up to 8 weeks post dose.
  Overall number of AEs, severity, and relationship to study treatment per treatment group.
Number of participants with abnormalities in any laboratory parameter | Part A: up to 12 weeks post dose. Part B: up to 8 weeks post dose
  Safety laboratory data (blood chemistry, hematology, coagulation, and urinalysis)

SECONDARY OUTCOMES:
Number of AEs | up to 48 weeks post dose
  Overall number of AEs, severity and relationship to study treatment per treatment group
Number of participants with abnormalities in any laboratory parameter | up to 48 weeks post dose
  Safety laboratory data (blood chemistry, hematology, coagulation, and urinalysis)
Plasma pharmacokinetics of QCZ484 and metabolites - Cmax | Day 1; up to Day 8
  Measured by Cmax - The maximum plasma concentration of QCZ484 and of potential metabolites
Plasma pharmacokinetics of QCZ484 - Tmax | Day 1; up to Day 8
  Measured by Tmax - Time to Reach the Maximum Concentration After Drug Administration of QCZ484
Plasma pharmacokinetics of QCZ484 and metabolites - AUC0-48 | Day 1; up to Day 8
  Measured by AUC - Area under the curve versus time curve of QCZ484 from 0 to 48 hours (AUC0-48) and of potential metabolites
Plasma pharmacokinetics of QCZ484 - AUC0-inf | Day 1; up to Day 8
  Measured by AUC - Area under the curve versus time curve of QCZ484 from 0 to infinity (AUC0-inf)
Plasma pharmacokinetics of QCZ484 - T1/2 | Day 1; up to Day 8
  Measured by T1/2 - The elimination half-life of QCZ484
Urine pharmacokinetics of QCZ484 | Day 1; up to Day 2
  Measured by urine concentration of QCZ484 up to 24 hours post dose
Change from baseline in serum angiotensinogen (AGT) level | up to 48 weeks post dose
  Measured by serum AGT level

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (3):
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Morayfield, Queensland
  - Novartis Investigative Site, Adelaide
- Novartis Investigative Site, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No